CLINICAL TRIAL: NCT06978686
Title: The Validity and Reliability of the Turkish Version of the Barriers to Being Active Quiz
Brief Title: The Validity and Reliability of the Turkish Version of the BBAQ
Status: Recruiting | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Emel Mete, Assistant Professor, PhD, Istanbul Medeniyet University
Other Study IDs: 2025/BBAQ
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-05

CONDITIONS: Health Knowledge, Attitudes, Practice; Physical Inactivity
Keywords: exercise; questionnaires; physical activity; validation study
MeSH Terms: conditions — Behavior; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteers: This group consists of healthy university students between the ages of 18 and 35 who voluntarily participate in the study.

SUMMARY:
The Barriers to Being Active Quiz (BBAQ) was originally developed in English to identify barriers to physical activity. This study aims to translate and cross-culturally adapt the BBAQ into Turkish (BBAQ-T) and evaluate its psychometric properties.

DETAILED DESCRIPTION:
The study involves the translation and cross-cultural adaptation of the BBAQ into Turkish and the assessment of its reliability and validity. A total of 210 healthy participants will be recruited. The adaptation process will follow a standardized back-translation method using two bilingual translators. A pilot study (n=15) will assess face validity, including linguistic clarity, conceptual relevance, and administration time. To evaluate test-retest reliability, participants will complete the BBAQ-T again within 5-7 days after the initial assessment. Internal consistency will be analyzed using Cronbach's alpha (α). Construct validity will be examined by correlating the BBAQ-T with the Turkish versions of the Self-Perceived Barriers for Physical Activity Questionnaire and the Short Form-12 (SF-12).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Ability to read and write in Turkish
* No visual or hearing impairments that would interfere with participation
* Ability to follow simple instructions
* Willingness to participate in the study

Exclusion Criteria:

* Diagnosis of rheumatological conditions that may limit physical activity and are characterized by chronic inflammation and/or joint deformities (e.g., rheumatoid arthritis, ankylosing spondylitis, systemic lupus erythematosus, psoriatic arthritis)
* Physical limitations due to neurological or orthopedic conditions (e.g., stroke, cerebral palsy, multiple sclerosis, limb amputation, or orthopedic surgery within the past six months)
* History of psychiatric disorders that may impair cognitive functioning (e.g., schizophrenia, bipolar disorder, severe depression, attention deficit hyperactivity disorder)
* Presence of any cognitive impairment

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The sample will consist of volunteer, healthy participants.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Barriers to Being Active Quiz | Baseline (First assessment)
  The Barriers to Being Active Quiz (BBAQ) is a 21-item questionnaire originally developed by the Centers for Disease Control and Prevention (CDC) to identify perceived barriers to physical activity. Items are rated on a 4-point Likert-type scale ranging from 0 (very unlikely) to 3 (very likely). The scale includes seven sub-dimensions: lack of time, social influences, lack of energy, lack of willpower, fear of injury, lack of skills, and lack of resources. A subscale score of 5 or higher indicates a significant barrier in that domain. In this study, the BBAQ will be translated and cross-culturally adapted into Turkish following standardized guidelines.

SECONDARY OUTCOMES:
Barriers to Being Active Quiz | Within a 5-to-7-day period after the first assessment (Second assessment)
  The Barriers to Being Active Quiz (BBAQ) is a 21-item questionnaire originally developed by the Centers for Disease Control and Prevention (CDC) to identify perceived barriers to physical activity. Items are rated on a 4-point Likert-type scale ranging from 0 (very unlikely) to 3 (very likely). The scale includes seven sub-dimensions: lack of time, social influences, lack of energy, lack of willpower, fear of injury, lack of skills, and lack of resources. A subscale score of 5 or higher indicates a significant barrier in that domain. In this study, the BBAQ will be translated and cross-culturally adapted into Turkish following standardized guidelines
Self-Perceived Barriers for Physical Activity Questionnaire | Baseline (First assessment)
  This self-report instrument evaluates individuals' perceived obstacles to physical activity across personal, social, and environmental domains. It has been validated in Turkish and is used in this study to assess the convergent validity of the BBAQ-T. Participants rate the degree to which each item is a barrier to their physical activity.
Short Form-12 | Baseline (First assessment)
  The SF-12 is a widely used instrument that assesses health-related quality of life. It provides two summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). The Turkish version has been validated and will be used to further support the construct validity of the BBAQ-T by evaluating correlations with general health status

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - İstanbul Medeniyet University, Kartal, Istanbul
  - Emel Mete, Maltepe, Istanbul

IPD SHARING:
Plan to Share IPD: No